CLINICAL TRIAL: NCT04439110
Title: MATCH Treatment Subprotocol Q: Ado-trastuzumab Emtansine in Patients With Tumors With HER2 Amplification (Except Breast and Gastric/Gastro-Esophageal Junction (GEJ) Adenocarcinomas)
Brief Title: Testing Ado-Trastuzumab Emtansine as a Potential Targeted Treatment in Cancers With HER2 Genetic Changes (MATCH-Subprotocol Q)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-02979; NCI-2020-02979 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Q (Other: ECOG-ACRIN Cancer Research Group); EAY131-Q (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (trastuzumab emtansine) (Experimental): Patients receive trastuzumab emtansine IV over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Trastuzumab Emtansine

INTERVENTIONS:
Biological: Trastuzumab Emtansine — Given IV
  Other Names: Ado Trastuzumab Emtansine; ADO-Trastuzumab Emtansine; Kadcyla; PRO 132365; PRO-132365; PRO132365; RO5304020; T-DM1; TDM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate

SUMMARY:
This phase II MATCH treatment trial identifies the effects of ado-trastuzumab emtansine in patients whose cancer has a genetic change called HER2 amplification. Ado-trastuzumab emtansine is a monoclonal antibody, called trastuzumab, linked to a chemotherapy drug called DM1. Trastuzumab is a form of "targeted therapy", because it works by attaching itself to specific molecules (receptors) on the surface of cancer cells, known as HER2 receptors and delivers DM1 to kill them. Researchers hope to learn if the study drug will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive trastuzumab emtansine intravenously (IV) over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients' tumor sample must have HER2 amplification > 7 based on targeted custom Ampliseq panel on the Ion Torrent Personal Genome Machine (PGM)
* Hemoglobin >= 9.0 g/dL (which may be reached by transfusion)
* Patients will be allowed if on anticoagulation (except warfarin and other coumarin derivatives) or on aspirin 81 mg by mouth daily. Additional monitoring while on anticoagulation will be based on institutional guidelines and/or physician discretion. However, patients will not be allowed if on long acting anti-platelet agents such as clopidogrel
* Patients must have an electrocardiogram (ECG) within 4 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must have echocardiography (ECHO) or nuclear study (multigated acquisition scan [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have a left ventricular ejection fraction (LVEF) < 50% to be eligible
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 7 months after completion of study

Exclusion Criteria:

* Patients with a diagnosis of breast cancer or gastric/gastroesophageal junction (GEJ) cancer will be excluded
* Patients must not have known hypersensitivity to ado-trastuzumab emtansine or compounds of similar chemical or biologic composition
* Patients with current peripheral neuropathy of grade 3 or greater (National Cancer Institute [NCI]-Common Toxicity Criteria [CTC], version 4.0) will be excluded

  * Neuropathy assessment and grade assignment will be based on history (location, duration, balance and gait, effect on activity of daily living [ADLs]) and physical exam
* Patient must not have had any of the prior therapies:

  * Food and Drug Administration (FDA) approved:

    * Trastuzumab
    * Pertuzumab
    * Ado-trastuzumab emtansine
  * Investigational:

    * Margetuximab
    * PF-05280014 (Pfizer, Trastuzumab Biosimilar)
    * CT-P6 (Celltrion, Trastuzumab Biosimilar)
    * ABP-980 (Amgen, Trastuzumab Biosimilar)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2019-03-09 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Komal Jhaveri, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Q was activated on August 12, 2015. A total of 58 patients were assigned to this arm after screening, all from screening cohort. Of the 58 patients, 38 patients were enrolled to arm Q between November 19, 2015 and March 20, 2017.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol Q, patients had to have a tumor ERBB2 copy number of >7.
Period: Overall Study
Arm/Group | Treatment (Trastuzumab Emtansine)
Started | 38
Eligible | 36
Completed (Treatment continued until disease progression or intolerability.) | 0
Not Completed | 38
Not completed — Ineligible | 2
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Disease proression | 25
Not completed — Withdrawal by Subject | 1
Not completed — Alternative therapy | 1
Not completed — Other complicating disease | 1
Not completed — Personal reasons | 1
Not completed — Still on treatment | 1

BASELINE CHARACTERISTICS:
Population: Patients who were eligible and received protocol treatment
Arm/Group | Treatment (Trastuzumab Emtansine)
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 64 [39 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 26
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among eligible and treated patients. Objective response rate is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. For each treatment arm, 90% two-sided binomial exact confidence interval will be calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 3 cycles for the first 33 cycles and every 4 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trastuzumab Emtansine)
Number analyzed (Participants) | 36
percentage of participants | 2 [1 to 16.5]

2. Secondary Outcome: 6 Months Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 3 cycles for the first 33 cycles and every 4 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trastuzumab Emtansine)
Number analyzed (Participants) | 36
percentage of participants | 23.6 [14.2 to 39.2]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Median PFS will be estimated using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: Patients who were eligible and received protocol treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Trastuzumab Emtansine)
Number analyzed (Participants) | 36
months | 3.1 [2.1 to 4.4]

ADVERSE EVENTS:
Time Frame: Assessed every 21 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Arm/Group | Treatment (Trastuzumab Emtansine)
All-Cause Mortality (participants affected / at risk) | 30/38
Serious Adverse Events (participants affected / at risk) | 12/38
Other Adverse Events (participants affected / at risk) | 29/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trastuzumab Emtansine) (N=38)
Anemia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Ileal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Investigations - Other, specify (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Blurred vision (Eye disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trastuzumab Emtansine) (N=38)
Anemia (Blood and lymphatic system disorders) | 9
Chills (General disorders) | 2
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 14
Fever (General disorders) | 3
Gait disturbance (General disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Allergic reaction (Immune system disorders) | 2
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 11
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT04439110/Prot_SAP_000.pdf